CLINICAL TRIAL: NCT06465355
Title: The Role of Swallowing An Air Bolus on Primary Esophageal Peristalsis
Brief Title: Effects of an Air Bolus on Primary Peristalsis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Reza Shaker, MD, Associate Provost for Clinical and Translational Research, Senior Associate Dean and Director of the Clinical and Translational Science Institute of SE WI, and the Joseph E. Geenen Professor and Chief of Gastroenterology and Hepatology, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO00035855
Record Dates: First submitted 2024-06-10; First posted 2024-06-18 (Actual); Last update posted 2025-04-28 (Actual); Status verified 2025-04

CONDITIONS: Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: In healthy adults, determine the correlation between the transmission of a bolus from the pharynx into the proximal esophagus and activating primary esophageal peristalsis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy adults (Other): Pharyngo-esophageal high resolution manometry with affixed single-lumen, end-hole catheter wherein one end of the single lumen catheter is in the pharynx and the other is connected to an external stopcock to vent or not vent the pharynx to atmosphere during twenty dry swallows (10 vented, 10 unvented).
  Interventions: Procedure: pharyngo-esophageal high-resolution manometry

INTERVENTIONS:
Procedure: pharyngo-esophageal high-resolution manometry — The high resolution manometry (HRM) catheter will be inserted through the more patent nares and positioned such that it covers the pharynx and the esophagus. Affixed to the high resolution catheter will be a single lumen, end-hole catheter (length: 90 cm, outside diameter: 1.58 mm) wherein the end hole of the tube will be secured at a fixed pharyngeal site on the HRM catheter and the other end of the tube will be connected to a stopcock so that the tube may be either open or closed to atmospheric pressure. 3. Study subjects will be asked to swallow their ambient saliva ten times with the stopcock open and ten times with the stopcock closed. There is a 30 second interval between swallows.

SUMMARY:
Understanding the correlation between the transmission of a bolus from the pharynx into the proximal esophagus and activating primary esophageal peristalsis.

DETAILED DESCRIPTION:
Study Procedures and Analyses

1. All the study subjects are required to be without oral food or fluid intake for at least 3 hours prior to the study
2. After application of local lidocaine, the high resolution manometry (HRM) catheter will be inserted through the more patent nares and positioned such that it covers the pharynx and the esophagus. Affixed to the high resolution catheter will be a single lumen, end-hole catheter (length: 90 cm, outside diameter: 1.58 mm) wherein the end hole of the tube will be secured at a fixed pharyngeal site on the HRM catheter and the other end of the tube will be connected to a stopcock so that the tube may be either open or closed to atmospheric pressure.
3. Study subjects will be asked to swallow their ambient saliva ten times with the stopcock open and ten times with the stopcock closed. There is a 30 second interval between swallows.
4. Following completion of the study, the manometry catheter and the single lumen tube will be removed.
5. The participant will also be instructed to resume their regular diet and activity.
6. All the pressure recordings will be analyzed by two individuals in a blinded fashion.

The investigators will compare motility pressure metrics like striated esophageal muscle contractile integral, esophageal smooth muscle contractile integral, peristaltic wave velocity and esophageal clearance time to evaluate the potential differences in esophageal motility metrics when an air bolus is allowed to flow into the esophagus compared to those metrics when air is shunted out of the pharynx by a trans-nasal tube vented to the atmosphere.

Statistical analysis will be performed in a repeated measures technique comparing metrics with and without the pharyngeal shunt stopcock closed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subject with no history or present diagnosis of pharyngo-esophageal diseases or motility disorders
* Age 21 to 90 years

Exclusion Criteria:

* Under the age of 21
* Over the age of 90
* Presence of pharyngo-esophageal disease or motility disorders
* Pregnancy
* Lidocaine allergy

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
striated esophageal muscle contractile integral | through study completion, an average of 1 year
  Motility pressure metric to measure contractile vigor of the proximal esophagus in mmHg-cm-seconds
smooth esophageal muscle contractile integral | through study completion, an average of 1 year
  Motility pressure metric to measure contractile vigor of the distal esophagus in mmHg-cm-seconds
peristaltic wave velocity | through study completion, an average of 1 year
  average speed at which the primary peristaltic pressure wave traverses the esophagus in cm/second
esophageal clearance time | through study completion, an average of 1 year
  time for the entire swallowed bolus to travers the esophagus in seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No